CLINICAL TRIAL: NCT02284568
Title: A Multinational, Multicenter, Randomized, Double Blind, Parallel Group, Placebo Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Once Daily Oral Administration of Laquinimod (0.6 or 1.5 mg) in Patients With Primary Progressive Multiple Sclerosis (PPMS)
Brief Title: A Phase 2 Clinical Study in Subjects With Primary Progressive Multiple Sclerosis to Assess the Efficacy, Safety and Tolerability of Two Oral Doses of Laquinimod Either of 0.6 mg/Day or 1.5mg/Day (Experimental Drug) as Compared to Placebo
Acronym: ARPEGGIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TV5600-CNS-20006; 2014-001579-30 (EudraCT Number)
Record Dates: First submitted 2014-10-31; First posted 2014-11-06 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Primary Progressive Multiple Sclerosis
Keywords: multiple sclerosis; primary progressive multiple sclerosis; oral immunomodulator
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): once daily oral dose
  Interventions: Drug: Placebo
- Laquinimod 0.6 mg (Experimental): 1 capsule containing 0.6 mg laquinimod and 2 capsules containing placebo were administered orally once daily for at least 48 weeks.
  Interventions: Drug: Laquinimod; Drug: Placebo
- Laquinimod 1.5 mg (Experimental): 3 capsules containing 0.5 mg laquinimod were administered orally once daily for at least 48 weeks. However this arm was discontinued as of 01 January 2016 and no participants reached the 48 week timeframe.
  Interventions: Drug: Laquinimod

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Laquinimod — Laquinimod capsules in 0.5 mg and 0.6 mg strengths
  Other Names: TV-5600
  Arms: Laquinimod 0.6 mg; Laquinimod 1.5 mg
Drug: Placebo — Placebo capsules
  Arms: Laquinimod 0.6 mg

SUMMARY:
This Phase 2 study is intended to serve as a proof of concept for potential treatment with laquinimod in patients with PPMS. The study is also aimed at evaluating 2 doses of laquinimod in this population.

DETAILED DESCRIPTION:
Due to serious cardiovascular adverse events, Data Monitoring Committee (DMC) made a recommendation to stop all laquinimod treatment arms above 0.6 mg in the multiple sclerosis (MS) trials; therefore the 1.5 mg treatment arm in the ARPEGGIO study was discontinued as of 01 January 2016.

The DMC did not identify any definite cardiovascular risk in the 0.6 mg treatment arm, but felt that long term monitoring for emergence of any potential signal was necessary. Therefore, the 0.6 mg treatment arm was continued while the sponsor closely monitored cardiovascular events in all laquinimod studies. Prior to 01 January 2016, eligible patients were randomized in a 1:1:1 ratio into 1 of the following treatment arms (a total of 286 patients were randomized 1:1:1 prior to

01 January 2016):

* Laquinimod 0.6 mg daily
* Laquinimod 1.5 mg daily
* Daily placebo

As of 01 January 2016, following the decision to discontinue the laquinimod 1.5 mg dose arm, additional eligible patients (87 patients) who were enrolled were randomized in a 1:1 ratio into one of the following treatment arms:

* Laquinimod 0.6 mg daily
* Daily placebo

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed and documented PPMS diagnosis as defined by the 2010 Revised McDonald criteria
2. Baseline magnetic resonance imaging (MRI) showing lesions consistent with PPMS in either or both brain and spinal cord
3. Patients must have an Expanded Disability Status Scale (EDSS) score of 3 to 6.5, inclusive, at both screening and baseline visits
4. Documented evidence of clinical disability progression in the 2 years prior to screening.
5. Functional System Score (FSS) of > or equal 2 for the pyramidal system or gait impairment due to lower extremity dysfunction
6. Patients must be between 25 to 55 years of age, inclusive
7. Women of child-bearing potential must practice an acceptable method of birth control for 30 days before taking the study drug, and 2 acceptable methods of birth control during all study duration and until 30 days after the last dose of treatment is administered.
8. Patients must sign and date a written informed consent prior to entering the study.
9. Patients must be willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

1. Patients with history of any multiple sclerosis (MS) exacerbations or relapses, including any episodes of optic neuritis.
2. Progressive neurological disorder other than PPMS.
3. Any MRI record showing presence of cervical cord compression.
4. Baseline MRI showing other findings (including lesions that are atypical for PPMS) that may explain the clinical signs and symptoms.
5. Relevant history of vitamin B12 deficiency.
6. Positive human T-lymphotropic virus Type I and II (HTLV-I/II) serology.
7. Use of experimental or investigational drugs in a clinical study within 24 weeks prior to baseline. Use of a currently marketed drug in a clinical study within 24 weeks prior to baseline would not be exclusionary, provided no other exclusion criteria are met.
8. Use of immunosuppressive agents, or cytotoxic agents, including cyclophosphamide and azathioprine within 48 weeks prior to baseline.
9. Previous treatment with fingolimod (GILENYA®, Novartis), dimethyl fumarate (TECFIDERA®, Biogen Idec Inc), glatiramer acetate (COPAXONE®, Teva), interferon-β (either 1a or 1b), intravenous immunoglobulin, or plasmapheresis within 8 weeks prior to baseline.
10. Use of teriflunomide (AUBAGIO®, Sanofi) within 2 years prior to baseline, except if active washout (with either cholestyramine or activated charcoal) was done 2 months or more prior to baseline.
11. Prior use of monoclonal antibodies ever, except for:

    1. natalizumab (TYSABRI®, Biogen Idec Inc), if given more than 24 weeks prior to baseline AND the patient is John Cunningham (JC) virus antibody test negative (as per medical history)
    2. rituximab, ocrelizumab, or ofatumumab, if B cell count (CD19, as per medical history) is higher than 80 cells/μL
12. Use of mitoxantrone (NOVANTRONE®, Immunex) within 5 years prior to screening. Use of mitoxantrone >5 years before screening is allowed in patients with normal ejection fraction and who did not exceed the total lifetime maximal dose.
13. Previous use of laquinimod.
14. Chronic (eg, more than 30 consecutive days or monthly dosing, with the intent of MS disease modification) systemic (intravenous, intramuscular or oral) corticosteroid treatment within 8 weeks prior to baseline.
15. Previous use of cladribine or alemtuzumab (LEMTRADA®, Sanofi).
16. Previous total body irradiation or total lymphoid irradiation.
17. Previous stem cell treatment, cell-based treatment, or bone marrow transplantation of any kind.
18. Patients who underwent endovascular treatment for chronic cerebrospinal venous insufficiency (CCSVI) within 12 weeks prior to baseline.
19. Use of moderate/strong inhibitors of cytochrome P450 (CYP) 3A4 within 2 weeks prior to baseline.
20. Use of inducers of CYP3A4 within 2 weeks prior to baseline.
21. Pregnancy or breastfeeding.
22. Serum levels ≥3× upper limit of the normal range (ULN) of either alanine aminotransferase (ALT) or aspartate aminotransferase (AST) at screening.
23. Serum direct bilirubin which is ≥2×ULN at screening.
24. Patients with a clinically significant or unstable medical or surgical condition that (in the opinion of the Investigator) would preclude safe and complete study participation, as determined by medical history, physical examinations, electrocardiogram (ECG), laboratory tests or chest X-ray.
25. A known history of hypersensitivity to gadolinium (Gd).
26. Glomerular filtration rate (GFR) < or equal 60 mL/min at screening visit.
27. Inability to successfully undergo MRI scanning, including claustrophobia.
28. Known drug hypersensitivity that would preclude administration of laquinimod, such as hypersensitivity to mannitol, meglumine or sodium stearyl fumarate.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (99):
- United States (15):
  - Teva Investigational Site 12966, Phoenix, Arizona
  - Teva Investigational Site 12967, Newport Beach, California
  - Teva Investigational Site 12962, San Francisco, California
  - Teva Investigational Site 12964, Aurora, Colorado
  - Teva Investigational Site 12973, Northbrook, Illinois
  - Teva Investigational Site 12975, Kansas City, Kansas
  - Teva Investigational Site 12969, Lenexa, Kansas
  - Teva Investigational Site 12977, Golden Valley, Minnesota
  - Teva Investigational Site 13010, Golden Valley, Minnesota
  - Teva Investigational Site 12965, Chesterfield, Missouri
  - Teva Investigational Site 12968, St Louis, Missouri
  - Teva Investigational Site 12963, New York, New York
  - Teva Investigational Site 12971, Charlotte, North Carolina
  - Teva Investigational Site 12976, Columbus, Ohio
  - Teva Investigational Site 12970, Uniontown, Ohio
- Canada (6):
  - Teva Investigational Site 11089, Calgary, AL
  - Teva Investigational Site 11084, Halifax, Nova Scotia
  - Teva Investigational Site 11081, Ottawa, Ontario
  - Teva Investigational Site 11087, Toronto, Ontario
  - Teva Investigational Site 11082, Montreal, Quebec
  - Teva Investigational Site 11088, Québec, Quebec
- Germany (15):
  - Teva Investigational Site 32505, Bad Mergentheim
  - Teva Investigational Site 32512, Bamberg
  - Teva Investigational Site 32510, Berlin
  - Teva Investigational Site 32522, Bochum
  - Teva Investigational Site 32509, Dresden
  - Teva Investigational Site 32517, Düsseldorf
  - Teva Investigational Site 32543, Goettigen
  - Teva Investigational Site 32514, Hamburg
  - Teva Investigational Site 32507, Hanover
  - Teva Investigational Site 32513, München
  - Teva Investigational Site 32504, München
  - Teva Investigational Site 32516, Rostock
  - Teva Investigational Site 32523, Trier
  - Teva Investigational Site 32503, Ulm
  - Teva Investigational Site 32511, Würzburg
- Italy (9):
  - Teva Investigational Site 30106, Cefalù
  - Teva Investigational Site 30110, Florence
  - Teva Investigational Site 30105, Gallarate
  - Teva Investigational Site 30108, Genova
  - Teva Investigational Site 30102, Milan
  - Teva Investigational Site 30107, Orbassano
  - Teva Investigational Site 30103, Padua
  - Teva Investigational Site 30101, Rome
  - Teva Investigational Site 30104, Rome
- Netherlands (3):
  - Teva Investigational Site 38068, Amsterdam
  - Teva Investigational Site 38067, Nijmegen
  - Teva Investigational Site 38069, Sittard
- Poland (10):
  - Teva Investigational Site 53262, Bialystok
  - Teva Investigational Site 53250, Bydgoszcz
  - Teva Investigational Site 53253, Gdansk
  - Teva Investigational Site 53257, Katowice
  - Teva Investigational Site 53258, Katowice
  - Teva Investigational Site 53256, Katowice
  - Teva Investigational Site 53255, Kielce
  - Teva Investigational Site 53260, Lublin
  - Teva Investigational Site 53261, Olsztyn
  - Teva Investigational Site 53252, Warsaw
- Russia (11):
  - Teva Investigational Site 50285, Kaluga
  - Teva Investigational Site 50288, Kazan'
  - Teva Investigational Site 50290, Kazan'
  - Teva Investigational Site 50294, Kirov
  - Teva Investigational Site 50292, Krasnoyarsk
  - Teva Investigational Site 50287, Moscow
  - Teva Investigational Site 50291, Nizhny Novgorod
  - Teva Investigational Site 50286, Novosibirsk
  - Teva Investigational Site 50295, Perm
  - Teva Investigational Site 50289, Saint Petersburg
  - Teva Investigational Site 50293, Saint Petersburg
- Spain (10):
  - Teva Investigational Site 31108, Barcelona
  - Teva Investigational Site 31106, Barcelona
  - Teva Investigational Site 31104, Donostia / San Sebastian
  - Teva Investigational Site 31105, El Palmar
  - Teva Investigational Site 31111, Lleida
  - Teva Investigational Site 31112, Madrid
  - Teva Investigational Site 31192, Madrid
  - Teva Investigational Site 31101, Málaga
  - Teva Investigational Site 31102, Seville
  - Teva Investigational Site 31100, Valencia
- Ukraine (10):
  - Teva Investigational Site 58158, Dnipropetrovsk
  - Teva Investigational Site 58159, Ivano-Frankivsk
  - Teva Investigational Site 58157, Kharkiv
  - Teva Investigational Site 58160, Kyiv
  - Teva Investigational Site 58152, Lutsk
  - Teva Investigational Site 58154, Lviv
  - Teva Investigational Site 58153, Lviv
  - Teva Investigational Site 58156, Zaporizhzhia
  - Teva Investigational Site 58150, Zaporizhzhya
  - Teva Investigational Site 58151, Zaporizhzhya
- United Kingdom (10):
  - Teva Investigational Site 34190, Bristol
  - Teva Investigational Site 34188, Edinburgh
  - Teva Investigational Site 34189, Exeter
  - Teva Investigational Site 34182, Liverpool
  - Teva Investigational Site 34181, London
  - Teva Investigational Site 34183, Nottingham
  - Teva Investigational Site 34184, Oxford
  - Teva Investigational Site 34186, Plymouth
  - Teva Investigational Site 34185, Stoke-on-Trent
  - Teva Investigational Site 34187, Swansea

REFERENCES:
- [Derived] Falet JR, Durso-Finley J, Nichyporuk B, Schroeter J, Bovis F, Sormani MP, Precup D, Arbel T, Arnold DL. Estimating individual treatment effect on disability progression in multiple sclerosis using deep learning. Nat Commun. 2022 Sep 26;13(1):5645. doi: 10.1038/s41467-022-33269-x. PMID 36163349
- [Derived] Giovannoni G, Knappertz V, Steinerman JR, Tansy AP, Li T, Krieger S, Uccelli A, Uitdehaag BMJ, Montalban X, Hartung HP, Pia Sormani M, Cree BAC, Lublin F, Barkhof F. A randomized, placebo-controlled, phase 2 trial of laquinimod in primary progressive multiple sclerosis. Neurology. 2020 Aug 25;95(8):e1027-e1040. doi: 10.1212/WNL.0000000000010284. Epub 2020 Jul 10. PMID 32651286

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 447 patients were screened for enrollment into this study. Of the patients screened, 374 patients met entry criteria and were enrolled into the study. One participant withdrew before taking any study drug.
Groups:
- Placebo: 3 capsules containing placebo were administered orally once daily for at least 48 weeks.
Period: Overall Study
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
Started | 140 (Intent to treat (ITT) population) | 139 (Intent to treat (ITT) population) | 95 (Intent to treat (ITT) population)
Safety Population | 140 | 138 | 95
Completed Week 48 MRI - on Treatment | 113 | 107 | 0
Completed | 109 | 93 | 0
Not Completed | 31 | 46 | 95
Not completed — Adverse Event | 2 | 9 | 4
Not completed — Withdrawal by Subject | 22 | 21 | 1
Not completed — Noncompliance with study drug admin | 1 | 2 | 0
Not completed — Noncompliance | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Sponsor requested patient stop treatment | 0 | 0 | 90
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Lack of Efficacy | 4 | 7 | 0
Not completed — Other | 1 | 2 | 0
Not completed — Withdrew before taking study drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg | Total
Number analyzed (Participants) | 140 | 139 | 95 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (7.18) | 46.1 (6.68) | 46.1 (7.21) | 46.3 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 57 | 45 | 169
  Male | 73 | 82 | 50 | 205
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 138 | 132 | 92 | 362
  Black | 0 | 2 | 2 | 4
  Asian | 0 | 2 | 0 | 2
  Other | 2 | 3 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not HIspanic or Latino | 135 | 134 | 91 | 360
  Hispanic or Latino | 4 | 5 | 1 | 10
  Unknown | 1 | 0 | 3 | 4
Weight [Mean (Standard Deviation); unit: kg] | 73.97 (16.809) | 75.91 (16.668) | 73.47 (14.831) | 74.57 (16.275)
Height [Mean (Standard Deviation); unit: cm] | 171.25 (9.818) | 172.61 (9.246) | 171.03 (9.677) | 171.70 (9.573)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.136 (5.0283) | 25.373 (4.5539) | 25.026 (4.1002) | 25.196 (4.6208)
Time Since First MS Symptom [Mean (Standard Deviation); unit: years] — Multiple sclerosis (MS)
  years | 7.4 (5.22) | 8.3 (6.33) | 8.5 (5.61) | 8.0 (5.76)
Time Since First PPMS Diagnosis [Mean (Standard Deviation); unit: years] — Primary progressive multiple sclerosis (PPMS)
  years | 3.1 (2.98) | 4.0 (4.05) | 4.1 (4.04) | 3.7 (3.70)
Normalized Brain Volume [Mean (Standard Deviation); unit: mL] — Obtained from magnetic resonance imaging (MRI) scans
  mL | 1457.9 (109.78) | 1461.3 (96.63) | 1455.2 (101.44) | 1458.5 (102.69)
Expanded Disability Status Scale (EDSS) [Count of Participants; unit: Participants] — EDSS is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The EDSS scale ranges from 0 to 10 in 0.5 unit increments with 0=no disability and 10=death due to MS. Only an Examining Neurologist administered the EDSS. The Examining Neurologist did not have access to the patient's medical records or source documents, including previous EDSS forms or adverse events.
  Participants
    EDSS score 3 | 10 | 12 | 10 | 32
    EDSS score 3.5 | 27 | 25 | 20 | 72
    EDSS score 4 | 24 | 30 | 18 | 72
    EDSS score 4.5 | 26 | 19 | 17 | 62
    EDSS score 5 | 17 | 15 | 6 | 38
    EDSS score 5.5 | 24 | 23 | 16 | 63
    EDSS score 6 | 9 | 12 | 4 | 25
    EDSS score 6.5 | 3 | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Brain Volume Change (PBVC) From Baseline to Week 48 Using a Repeated Measures ANCOVA Model
Description: Brain atrophy (BA) was measured using magnetic resonance imaging (MRI) scans of the brain. BA was analyzed using baseline-adjusted repeated measures analysis of covariance (ANCOVA- SAS® PROC MIXED) in which 1 contrast was constructed in order to compare between laquinimod 0.6 mg and placebo. The statistical model was a repeated measures analysis of covariance with treatment group, week, treatment group by week interaction, normalized brain volume at baseline, natural logarithm of T2 lesion volume at baseline, and country as fixed effects. Only on-treatment observations (include all the assessments done up to one month after the last dose of the study drug) were included. Values are adjusted means. The cancelled laquinimod 1.5 mg treatment arm was not included in the repeated measures ANCOVA model analysis. However PBVC by visit data are offered in outcome #2.
Time Frame: Baseline (at least 14 days but not more than 6 weeks prior to Day 1), Weeks 24, 48 and including early termination visits
Population: Modified Intent to Treat 1 (mITT1) population with at least 1 post-baseline PBVC value and will include assessments taken up to/including early termination/study completion visit.
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 128 | 124 | 0
percentage change from baseline | -0.454 (0.0897) | -0.438 (0.0945) |
Statistical Analysis 1: Comparison: Placebo vs Laquinimod 0.6 mg; The statistical model was a repeated measures analysis of covariance with treatment group, week, treatment group by week interaction, normalized brain volume at baseline, natural logarithm of T2 lesion volume at baseline, and country as fixed effects; Test type: Superiority; p = 0.903, Repeated Measures ANCOVA — significance at 0.05; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.2390 to 0.2705], Standard Error of Mean 0.1293

2. Primary Outcome: Percent Brain Volume Change (PBVC) From Baseline to Weeks 24 and 48
Description: Brain atrophy (BA) was measured using magnetic resonance imaging (MRI) scans of the brain. Early termination scans of participants who discontinued the study after week 36 are considered scans at week 48.
Time Frame: Baseline (at least 14 days but not more than 6 weeks prior to Day 1), Weeks 24, 48
Population: Modified Intent to Treat 1 (mITT1) population with at least 1 post-baseline PBVC value.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 131 | 128 | 47
percentage change from baseline
  Week 24: number analyzed (Participants) | 124 | 121 | 20
  Week 24 | -0.241 (0.8978) | -0.042 (0.7537) | -0.820 (1.2693)
  Week 48: number analyzed (Participants) | 114 | 110 | 1
  Week 48 | -0.455 (0.9770) | -0.418 (0.9806) | 0.550

3. Secondary Outcome: Percentage of Participants With 12-Week Confirmed Disability Progression (CDP) As Measured by Expanded Disability Status Scale (EDSS) up to Week 48
Description: CDP was defined as increase in EDSS of >=1 point from baseline EDSS, if EDSS at entry is ≤5.0 or increase of >=0.5 point, if EDSS at entry is >=5.5. This increase should be confirmed after at least 12 weeks. Progression cannot be confirmed during a protocol defined relapse. EDSS is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The EDSS scale ranges from 0 to 10 in 0.5 unit increments with 0=no disability and 10=death due to MS. Only an Examining Neurologist administered the EDSS. The Examining Neurologist did not have access to the patient's medical records or source documents, including previous EDSS forms or adverse events. If a patient died due to MS disease progression, the patient was analyzed as having CDP with the time to CDP as the onset date of progression. If a patient died due to MS before having progression, then the time to disability progression was censored using the date of death.
Time Frame: Baseline (Week 0), Weeks 12, 24, 36, 48 (end if treatment if < 48 weeks)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 140 | 139 | 95
percentage of participants | 23 | 17 | 1
Statistical Analysis 1: Comparison: Placebo vs Laquinimod 0.6 mg; The statistical model was a Cox proportional hazards regression model with treatment group, categorical EDSS at baseline (≤4.5 or >4.5), age at baseline, natural logarithm of T2 lesion volume at baseline, and country as fixed effects; Test type: Superiority; p = 0.426, Log Rank — significance at 0.05. p-value was from a log-rank test, and estimate and confidence limits were from a Cox model with treatment group as fixed effect, due to the violation of the proportionality assumption; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.48 to 1.37] — Laquinimod 0.6 mg vs placebo

4. Secondary Outcome: Percentage of Participants With 12-Week Confirmed Disability Progression (CDP) As Measured by Expanded Disability Status Scale (EDSS) or the Timed 25-foot Walk (T25FW) Test up to Week 48
Description: CDP was defined as
  increase in EDSS of >=1 point from baseline EDSS, if EDSS at entry is ≤5.0 or increase of >=0.5 point, if EDSS at entry is >=5.5 confirmed after at least 12 weeks, OR increase of >= 20% from baseline in the T25FW test, confirmed after at least 12 weeks.
  EDSS quantifies disability in MS and monitors changes in the level of disability over time. The EDSS scale is 0-10 in 0.5 unit increments with 0=no disability and 10=death due to MS. The T25-FW is a quantitative mobility and leg function performance test based on the average time of two trials in which participants walk 25 feet as quickly as possible. Increasing time scores indicate increasing impairment.
  If a patient died due to MS disease progression, the patient was analyzed as having CDP with the time to CDP as the onset date of progression. If a patient died due to MS before having progression, then the time to disability progression was censored using the date of death.
Time Frame: Baseline (Week 0), Weeks 12, 24, 36, 48 (end if treatment if < 48 weeks)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 140 | 139 | 95
percentage of participants | 34 | 32 | 2
Statistical Analysis 1: Comparison: Placebo vs Laquinimod 0.6 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.867, Regression, Cox — significance at 0.05; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.68 to 1.59] — Laquinimod 0.6 mg vs placebo

5. Secondary Outcome: Change From Baseline for the Timed 25-foot Walk (T25FW) Score at Weeks 12, 24, 36 and 48
Description: The T25FW is a quantitative mobility and leg function performance test based on the average time of two trials in which participants walk 25 feet as quickly as possible. In cases when a patient could not complete a T25FW trial due to the physical limitations, a value of 180 seconds was assigned for that trial (this is the maximal possible value for the T25FW test). Increasing time scores indicate increasing impairment. Baseline values are summaries of observed values. Week values are change from baseline values.
Time Frame: Baseline (Week 0), Weeks 12, 24, 36, 48
Population: Modified Intent to Treat #2 (mITT2) population is a subset of the ITT population. It includes all participants in the ITT population with at least 1 post baseline efficacy assessment other than PBVC.
Measure: Median (Full Range); unit: seconds
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 139 | 137 | 89
seconds
  Baseline | 7.750 [3.15 to 46.00] | 7.600 [4.20 to 88.40] | 6.850 [4.25 to 62.00]
  Week 12: number analyzed (Participants) | 135 | 130 | 55
  Week 12 | 0.100 [-8.85 to 16.00] | 0.050 [-56.90 to 113.05] | 0.100 [-6.15 to 172.00]
  Week 24: number analyzed (Participants) | 133 | 127 | 25
  Week 24 | 0.100 [-20.50 to 16.85] | 0.350 [-58.50 to 113.05] | 0.150 [-4.00 to 172.15]
  Week 36: number analyzed (Participants) | 123 | 118 | 4
  Week 36 | 0.200 [-18.15 to 21.80] | 0.450 [-64.60 to 113.05] | 12.550 [1.65 to 27.60]
  Week 48: number analyzed (Participants) | 121 | 108 | 0
  Week 48 | 0.300 [-22.65 to 134.00] | 0.050 [-63.50 to 68.35] |
Statistical Analysis 1: Comparison: Placebo vs Laquinimod 0.6 mg; placebo n=121 Laquinimod 0.6 mg n=108 The estimate of parameter, standard error, and 95% confidence intervals for change from baseline was from a Mann-Whitney-Wilcoxon Test using Hodges-Lehmann estimates; Test type: Superiority; p = 0.248, Repeated Measures ANCOVA — significance at 0.05. The p-value for ranked change from baseline values was from a repeated measures analysis of covariance with trt group, week, treatment group by week interaction, rank of T25FW score at baseline, and country as fixed effects; Mean Difference (Final Values) = -0.325, 95% CI 2-sided [-0.8500 to 0.2000], Standard Error of Mean 0.2679 — Laquinimod 0.6 mg vs. placebo treatment effect

6. Secondary Outcome: Number of New T2 Brain Lesions at Week 48
Description: Inflammatory disease activity was assessed by magnetic resonance imaging (MRI) measurement of the number of new T2 lesions at week 48 as compared to baseline. Scans of patients who discontinued the study after week 36 are considered scans at week 48, and are included in week 48.
Time Frame: Baseline (Week 0), 48 weeks
Population: Modified intent to treat 1 (mITT1) population includes participants with at least 1 post-baseline PBVC value. Participants from the mITT1 with MRI data at week 48 are reported .
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 119 | 112 | 1
lesions | 3.5 (10.82) | 1.3 (3.01) | 1.0
Statistical Analysis 1: Comparison: Placebo vs Laquinimod 0.6 mg; This analysis was performed using baseline adjusted negative binomial regression model (SAS® PROC GENMOD) in which 1 contrast for comparing laquinimod 0.6 mg to placebo was constructed. In addition to the treatment group, the natural logarithm of T2 lesion volume at baseline, age at baseline and country/geographical region (CGR) were used as covariates; Test type: Superiority; p = 0.001, negative binomial regression model — significance at 0.05; Risk Ratio (RR) = 0.4, 95% CI 2-sided [0.26 to 0.69], Standard Error of Mean 0.11 — Laquinimod 0.6 mg vs. placebo risk ratio

7. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents usual activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 up to Week 130 (longest duration of treatment)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 140 | 138 | 95
Participants
  Any TEAE | 109 | 115 | 63
  Severe TEAE | 6 | 6 | 3
  Treatment-related TEAE | 27 | 41 | 29
  Deaths | 0 | 0 | 1
  Serious TEAE | 6 | 10 | 3
  Withdrawn from treatment due to TEAE | 2 | 8 | 4

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 130 (longest duration of treatment)
Arm/Group | Placebo | Laquinimod 0.6 mg | Laquinimod 1.5 mg
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/138 | 1/95
Serious Adverse Events (participants affected / at risk) | 6/140 | 10/138 | 3/95
Other Adverse Events (participants affected / at risk) | 77/140 | 74/138 | 40/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=140) | Laquinimod 0.6 mg (N=138) | Laquinimod 1.5 mg (N=95)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Testicular abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HIV test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbosacral plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=140) | Laquinimod 0.6 mg (N=138) | Laquinimod 1.5 mg (N=95)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 5 (5) | 5 (5)
Constipation (Gastrointestinal disorders) | 6 (8) | 7 (7) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 9 (12) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 6 (6)
Fatigue (General disorders) | 5 (5) | 7 (7) | 3 (3)
Influenza (Infections and infestations) | 13 (15) | 7 (7) | 2 (2)
Nasopharyngitis (Infections and infestations) | 24 (31) | 24 (34) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 12 (16) | 2 (2)
Urinary tract infection (Infections and infestations) | 11 (16) | 9 (13) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 9 (13) | 9 (15) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (10) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 12 (15) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6) | 1 (2)
Headache (Nervous system disorders) | 16 (28) | 14 (16) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT02284568/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT02284568/SAP_001.pdf